CLINICAL TRIAL: NCT07317856
Title: Efficacy of Microneedling With Hyaluronic Acid Injection for Gingival Augmentation in Thin Gingival Phenotype: A Split- Mouth Randomized Clinical Trial
Brief Title: Efficacy of Microneedling With Hyaluronic Acid Injection for Gingival Augmentation in Thin Gingival Phenotype
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Murtadha Muhammed Humadi, Dentist, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1114
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Thin Gingival Biotype
Keywords: Hyaluronic acid; microneedling; soft tissue regeneration; soft tissue augmentation
MeSH Terms: interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Intervention Model Description: The study will be a 6-month follow-up, split mouth, double blind, prospective randomized controlled Clinical trial
Who Masked: Outcomes Assessor
Masking Description: A double-blind design is implemented where both the outcome assessor and the statistician responsible for data analysis remain blinded to treatment allocation throughout the study. The outcome assessor, who is a calibrated examiner does not present during intervention procedures, performs all clinical measurements without knowledge of the interventions received at each site. Clinical measurements and standardized intraoral photographs are coded using an anonymous site numbering system without reference to actual treatments received. Similarly, the statistician remains blinded to treatment codes until completion of the final statistical analysis, with treatment groups coded using anonymous identifiers throughout data collection and analysis phases to prevent analytical bias
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microneedling (MN) Group (Active Comparator): Control group
  Interventions: Procedure: Microneedling (MN)
- Microneedling + Injectable Hyaluronic Acid (MN + HA) Group (Experimental): Test group
  Interventions: Combination Product: Microneedling + Injectable Hyaluronic Acid (MN + HA)

INTERVENTIONS:
Procedure: Microneedling (MN) — A derma pen (Dr. Pen Ultima A6) with 24-pin cartridge will be used for microneedling. The device will be vertically inserted through the keratinized gingiva at each treatment site until contact with the underlying hard tissue (bone) is reached. Treatment will extend from the mesial line angle of the central incisor to the distal line angle of the canine. The treatment endpoint is identified as uniform pin-point bleeding, which is easily controlled with gentle pressure. The microneedling procedure will be repeated for three sessions, with each session spaced 7 days apart. This protocol ensures consistent intervention dosage and timing to optimize gingival augmentation outcomes while allowing adequate healing time between sessions.
  Arms: Microneedling (MN) Group
Combination Product: Microneedling + Injectable Hyaluronic Acid (MN + HA) — A derma pen (Dr. Pen Ultima A6) with 24-pin cartridge will be used for microneedling. The device will be vertically inserted through the keratinized gingiva at each treatment site until contact with the underlying hard tissue (bone) is reached. Treatment will extend from the mesial line angle of the central incisor to the distal line angle of the canine.The hyaluronic acid injection protocol for gingival augmentation utilizes cross-linked hyaluronic acid at 16-20 mg/mL concentration with 200-400 μm particle size, delivered via sterile pre-filled syringes using 30-gauge microneedles (8mm) with 1mL insulin syringes marked at 0.02mL intervals. Following topical anesthetic application for 2-3 minutes, the injection technique targets two anatomical sites per treatment area: the first point located 3mm apical to the free gingival margin and the second point apical to the mucogingival junction. Post-injection gentle circular massage for 2-3 minutes ensures uniform distribution of the material
  Arms: Microneedling + Injectable Hyaluronic Acid (MN + HA) Group

SUMMARY:
This randomized controlled trial adheres to the Consolidated Standards of Reporting Trials (CONSORT) 2010 guidelines and the Declaration of Helsinki ethical principles for medical research. The study complies with Good Clinical Practice (GCP) standards and will be prospectively registered with ClinicalTrials.gov to ensure transparency and accountability. A crossover design is implemented to ensure all participants receive both treatment modalities-microneedling (MN) alone and microneedling combined with injectable hyaluronic acid (MN + HA)-following an appropriate washout period, promoting equitable access while maintaining scientific rigor through within-subject comparisons.

Baseline Preparation

All enrolled participants receive comprehensive periodontal therapy at baseline, including supragingival and subgingival scaling using ultrasonic instrumentation combined with hand instruments. Standardized oral hygiene protocols are established with identical oral care products provided to each subject, including a soft-bristled toothbrush and interdental cleaning aids. All participants receive instruction in proper brushing technique with emphasis on twice-daily maintenance to ensure consistent plaque control throughout the trial.

Microneedling Intervention

The MN intervention comprises three sessions spaced seven days apart. Following baseline clinical assessment (plaque index, bleeding on probing, probing depth, clinical attachment level, keratinized tissue width, and gingival thickness) with standardized photographs, topical anesthesia is applied for one minute followed by infiltration anesthesia with 2% lidocaine with 1:100,000 epinephrine. The Dr. Pen Ultima A6 with a 24-pin cartridge is vertically inserted through keratinized gingiva until bone contact is achieved, treating from the mesial central incisor to the distal canine. Treatment ends when uniform pin-point bleeding is achieved. Post-procedure care includes gentle saline rinse, avoidance of brushing for 24 hours, twice-daily 0.12% chlorhexidine mouthwash for seven days, and avoidance of NSAIDs. Clinical reassessment occurs at 3 and 6 months.

Microneedling Plus Hyaluronic Acid Intervention

Following identical baseline assessment, anesthesia, and microneedling as the MN group, cross-linked hyaluronic acid (16-20 mg/mL, 200-400 µm particle size) is injected using 30-gauge needles (8 mm) with 1 mL insulin syringes. Two anatomical sites per area receive injections: 3 mm apical to the free gingival margin and apical to the mucogingival junction. The needle is inserted at 45 degrees, advanced 2-3 mm until blanching occurs, with a total volume of 0.04 mL per site (0.02 mL per point) at a rate not exceeding 0.01 mL per 10 seconds. Post-injection circular massage for 2-3 minutes ensures uniform distribution. Three sessions are performed seven days apart with identical post-procedure care and follow-up assessments at 3 and 6 months.

Outcome Measures

The primary outcome is the change in gingival thickness (millimeters) at treated sites from baseline to 6 months post-intervention, measured using transgingival probing. Secondary outcomes include changes in keratinized gingiva width, periodontal parameters (Plaque Index, Bleeding on Probing, Probing Pocket Depth, and Clinical Attachment Level), and patient-reported outcomes for pain, swelling, discomfort, and bleeding measured using visual analog scales at 2, 24, and 48 hours post-intervention. This comprehensive protocol ensures robust evaluation of both objective tissue augmentation and subjective patient experiences across both treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years from both sexes
* Systemically healthy individuals with no history of chronic systemic diseases.
* Participants with positive periodontal probe transparency in anterior teeth.
* Adequate oral hygiene (full-mouth plaque score ≤20%).
* Non-smokers or former smokers who quit ≥12 months prior to enrollment.
* Willingness to comply with study procedures, attend follow-up visits, and provide written informed consent.

Exclusion Criteria:

* Pregnancy or lactation.
* Use of medications affecting periodontal status or wound healing (e.g., systemic corticosteroids, bisphosphonates) within the past six months
* History of periodontal surgery or soft-tissue augmentation procedures at the target sites
* Active periodontal disease (probing depth >3 mm, clinical attachment loss >2 mm) or gingival inflammation (bleeding on probing ≥ 10%).
* Untreated carious lesions or periapical pathology in the study area.
* Systemic conditions that impair healing (e.g., uncontrolled diabetes mellitus, immunocompromised states).
* Use of anti-inflammatory or anticoagulant medications within two weeks prior to treatment.
* Known allergy to hyaluronic acid or components of the microneedling device.
* Presence of heavy gingival pigmentation at the target sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in gingival thickness | 6 months
  The primary outcome measure is the change in gingival thickness (in millimeters) at treated sites from baseline to 6 months post-intervention, as determined by transgingival probing method.

SECONDARY OUTCOMES:
Change in width of keratinized gingiva | 6 months
Plaque Index (PI) | 6 months
Bleeding on probing (BOP) | 6 months
Clinical attachment level (CAL) | 6 months
Change in probing depth | 6 months
Patient-reported outcomes | 48 hours
  Patient-reported outcomes assessed via visual analog scales for pain, swelling, discomfort and bleeding at 2 hours, 8 hours, 24 hours, and 48 hours following each intervention session.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided